CLINICAL TRIAL: NCT06322342
Title: A Multi-Center, Phase 2, Open Label, Ascending Dose Study to Evaluate the Safety and Efficacy of RVP-001 and to Identify an Appropriate Dose to Detect CNS Lesions in Adult Patients
Brief Title: Phase 2 Ascending Dose Safety and Efficacy Study of RVP-001, a Manganese-based MRI Contrast Agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reveal Pharmaceuticals Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: RVL-102-23; 9R44CA261240-04A1 (NIH)
Record Dates: First submitted 2024-03-11; First posted 2024-03-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Central Nervous System (CNS) Lesions; Brain Metastases; Brain Neoplasms; Brain Neoplasms, Benign; Brain Tumor, Primary; Brain Tumor, Recurrent; Brain Tumors; Brain Cancer; Brain Tumor; Brain Neoplasm, Primary; Multiple Sclerosis; Multiple Sclerosis Brain Lesion; Neurofibroma; Acoustic Neuroma; CNS Tumor; CNS Lesion; CNS Metastases; CNS Cancer; CNS Lymphoma; Von Hippel Lindau; Meningioma; Glioma; Schwannomas; Neuroinflammation; Neoplasia
MeSH Terms: conditions — Brain Neoplasms; Multiple Sclerosis; Neurofibroma; Neuroma, Acoustic; Central Nervous System Neoplasms; Meningioma; Glioma; Neurilemmoma; Neuroinflammatory Diseases; Neoplasms | interventions — Mn-PyC3A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 mg/Mn/kg (Experimental): 6 subjects each will receive RVP-001 at a dose of 2 mg Mn/kg
  Interventions: Drug: RVP-001
- 7 mg/Mn/kg (Experimental): 6 subjects each will receive RVP-001 at a dose of 7 mg Mn/kg
  Interventions: Drug: RVP-001
- 12 mg/Mn/kg (Experimental): 6 subjects each will receive RVP-001 at a dose of 12 mg Mn/kg
  Interventions: Drug: RVP-001

INTERVENTIONS:
Drug: RVP-001 — MRI contrast agent
  Other Names: Mn-PyC3A; mangaverate

SUMMARY:
This Phase 2 clinical trial will study RVP-001, a new manganese-based MRI contrast agent, in people who are known to have gadolinium-enhancing central nervous system (CNS) lesions, for example brain tumors or multiple sclerosis.

The goal of this study is to assess safety, efficacy, and pharmacokinetics of RVP-001 at three dose levels. The study will also compare RVP-001 imaging to gadolinium-based contrast agent (GBCA) imaging. A single dose of RVP-001 will be administered to each subject. Subjects will have known gadolinium-enhancing CNS lesions and will have a gadolinium-based contrast agent-enhanced MRI of the brain 2-14 days before receiving RVP-001 with imaging.

The ultimate goal of this research program is development of a gadolinium-free alternative to current general purpose MRI contrast agents.

DETAILED DESCRIPTION:
Subjects may include individuals who have a stable primary brain tumor, metastatic brain tumors, multiple sclerosis, or other gadolinium-enhancing CNS lesions. Following the screening GBCA-enhanced MRI scan to confirm presence of target lesion(s), a baseline unenhanced MRI scan will be performed prior to RVP-001 injection. Dynamic imaging will be performed in conjunction with RVP-001 injection. Steady state imaging will follow at multiple time points during the first hour following dose administration to characterize the pharmacodynamics of RVP-001 and to assess its ability to enhance visualization of areas with disrupted blood brain barrier and/or abnormal vascularity of the central nervous system.

Three dose cohorts are planned.

An unenhanced MRI scan follow-up study will be performed between one week and six weeks following the administration of RVP-001.

Safety will be evaluated throughout the study by assessing the following parameters: adverse events (AEs), physical examinations, injection site monitoring, electrocardiograms (ECGs), vital signs, clinical laboratory evaluations, medical history, and prior and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of all sexes, aged 18-75 years
2. Patients with known enhancing CNS lesions, including but not limited to gliomas, meningiomas, glioblastomas, schwannomas, brain metastases, multiple sclerosis lesions, that are on an ongoing follow-up MRI schedule
3. Patients who have had a GBCA-enhanced MRI within the past 14 days which demonstrated focal areas of disrupted Blood Brain Barrier (BBB) (e.g., primary and secondary tumors, focal inflammatory disorders) including at least one enhancing lesion of minimum 5 mm (long axis)
4. Acceptable renal function

Exclusion Criteria:

1. Serious non-malignant disease that could compromise protocol objectives in the opinion of the investigator and/or the Sponsor
2. Body mass index (BMI) greater than 35
3. Patients with clinically significant cardiac disease
4. MRI incompatibility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From time of dosing to 7 days post dose
  Treatment-emergent adverse events for each dose level will be summarized.
Lesion visualization criteria for RVP-001 enhanced MRI compared to unenhanced MRI | 1 day
  The lesion visualization criteria is based on 3 criteria: border delineation, lesion contrast, and internal morphology. These criteria will be assessed by independent readers for representative lesions using the images acquired during the MRI performed with RVP-001.
Lesion visualization criteria for RVP-001 compared to gadolinium-based contrast agent (GBCA) | 1 day
  The lesion visualization criteria is based on 3 criteria: border delineation, lesion contrast, and internal morphology. These criteria will be assessed by independent readers for representative lesions using the images acquired with RVP-001 and those acquired with the GBCA.
  For each reader, only matching lesion-pairs present in both MRI image sets (using GBCA and RVP-001) will be considered.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No